CLINICAL TRIAL: NCT01801787
Title: The Mechanism of Non-invasive Brain Stimulation for Therapy of Chronic Auditory Verbal Hallucinations in Schizophrenia
Brief Title: Non-invasive Brain Stimulation for Auditory Verbal Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andres Neuhaus, MD, M.D., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EA4/123/12
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Auditory Verbal Hallucinations; Schizophrenia
MeSH Terms: conditions — Hallucinations; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- verum tDCS (Experimental): left-hemispheric tDCS: anode placed midway between F3 and FP1, cathode placed midway between T3 and P3
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): left-hemispheric sham tDCS: anode placed midway between F3 and FP1, cathode placed midway between T3 and P3
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — active vs. sham tDCS left hemisphere
  Other Names: device: neuroConn tDCS PLUS device

SUMMARY:
The current study investigates the basic principles that underlie the efficacy of transcranial direct current stimulation for chronic auditory verbal hallucinations in schizophrenia in a multimodal design.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia
* chronic auditory verbal hallucinations
* right-handed

Exclusion Criteria:

* drug abuse other than nicotine
* severe cognitive deficits
* severe medical conditions
* severe neurological disorders
* severe microangiopathy
* history of electroconvulsive therapy
* pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of Auditory Hallucination Rating Scale score | baseline; 3 days after intervention; 3 months after intervention
  Auditory Hallucination Rating Scale score will be assessed at baseline; changes thereof at 3 days after intervention and 3 months after intervention are primary outcome measures

SECONDARY OUTCOMES:
Positive And Negative Syndrome Scale | baseline; 3 days after intervention; 3 months after intervention
  Positive And Negative Syndrome Scale score will be assessed at baseline; changes thereof at 3 days after intervention and 3 months after intervention are secondary outcome measures

OTHER OUTCOMES:
N1 suppression during talking and listening | baseline; 3 days after intervention
  N1 suppression during talking and listening will be assessed at baseline; change thereof at 3 days after intervention is further outcome measure
Diffusion Tensor Imaging: Fractional anisotropy of longitudinal superior fascicle and arcuate fascicle | baseline; 3 days after intervention
  Fractional anisotropy of longitudinal superior fascicle and arcuate fascicle will be assessed at baseline; change thereof 3 days after intervention is further outcome measure
Default Mode Network connectivity | baseline; 3 days after intervention
  Default Mode Network connectivity will be assessed at baseline; change thereof 3 days after intervention is further outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lindenberg, MD, Principal Investigator — Department of Neurology, Charité University Medicine Berlin; Andres H. Neuhaus, MD, Principal Investigator — Department of Psychiatry, Charité University Medicine Berlin
Locations (1):
- Charité University Medicine, Berlin, Germany